CLINICAL TRIAL: NCT01741740
Title: High Incidence of Chronic Complaints and Recurrence 5 Years After Simple Sutured Umbilical Hernia Repair
Brief Title: Chronic Complaints After Small Umbilical Hernia Repair
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Thue Bisgaard, MD, DMSc, Hvidovre University Hospital
Other Study IDs: SMALLUMBI123
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Chronic Pain; Ventral Hernia
Keywords: pain, hernia, chronic, discomfort, retrospective
MeSH Terms: conditions — Chronic Pain; Hernia, Ventral; Pain; Hernia; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- retrospective surgical patients: consecutive elective umbilical hernia repair patients during two years from two hospitals,- retrospective id with prospective follow up

SUMMARY:
There are only little data on the risk of chronic complaints (pain and discomfort) following open non-mesh sutured repairs of small umbilical or epigastric hernias. Our primary and secondary endpoints were long-term pain and discomfort at rest, respectively and thirdly recurrence. The setup was a retrospective two-centre study including patients ≥18 years undergoing primary elective open non-mesh sutured umbilical or epigastric hernia repairs. The survey included questions on suspicion of recurrence, reoperation for recurrence (if yes patients were examined by a consultant in patients home), pain, discomfort, work, and leisure activities. We analysed 295 consecutive patients through a non-validated structured questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* primary elective open non-mesh sutured umbilical or epigastric hernia repair

Exclusion Criteria:

* mesh repair, acute repair, repair secondary to other operation, recurrent hernia repair, combined hernia repair, laparoscopic hernie repair, trocar hernia repair, incompensated liver cirrhosis, age < 18 years, pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing primary elective open non-mesh sutured umbilical or epigastric hernia repair during a five years period
Sampling Method: Non-Probability Sample
Enrollment: 295 (Actual)
Dates: Start 2000-01; Primary Completion 2005-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
pain at rest at the hernia repair site | chronic complaints 5 years after hernia repair
  a verbal rating scale for pain is used (none, little, moderate or severe

SECONDARY OUTCOMES:
discomfort at rest at the hernia site | 5 years
  a verbal rating scale for pain is used (none, little, moderate or severea

OTHER OUTCOMES:
recurrence | five years
  reoperation for recurrence combined with clinical examination for non reoperated recurrences

CONTACTS AND LOCATIONS:
Overall Officials: Thue Bisgaard, DMSc, Principal Investigator — Hvidovre and Glostrup University Hospitals